CLINICAL TRIAL: NCT01174953
Title: High Risk Prostate Cancer Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12052
Record Dates: First submitted 2010-07-26; First posted 2010-08-04 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Finasteride plus soy (Other): Finasteride and soy
  Interventions: Drug: finasteride

INTERVENTIONS:
Drug: finasteride — Finasteride 5 mg once daily
  Soy 4 capsules twice daily (160 mg total)
  Other Names: Proscar; Propecia; isolavone

SUMMARY:
The purpose of this study is to study the molecular effects of the chemopreventative agent, finasteride, in combination with dietary soy supplementation in patients at high risk for the development of prostate cancer. Also, the investigators intend to create a large database with health information from men who are at high risk of developing prostate cancer, along with serum and tissue samples from those patients who are willing to provide tissue and serum samples.

DETAILED DESCRIPTION:
Over 180,000 new cases of prostate cancer are diagnosed in the United States each year, making prostate cancer the most frequently diagnosed cancer in men. With an estimated 28,660 deaths occurring in 2008, prostate cancer is the second leading cause of cancer death in men. In Kansas, prostate cancer is also the most frequent cancer among men and ranked third (253 deaths in 2006) behind lung cancer (884 deaths in 2006) and colorectal cancer (273 deaths in 2006) in cancer related mortality. Despite the significant morbidity and mortality related to this disease, screening and treatment approaches remain controversial and there is significant morbidity related to the treatment of early stage disease. Preventative strategies and strategies which identify patients at highest risk are needed desperately.

The goal of this proposal is to study the molecular effects of the chemopreventative agent, finasteride in combination with dietary soy supplementation in patients at high risk for the development prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Based on the PSA, DRE and Family history of prostate cancer patients will be risk stratified using Prostate Cancer Risk Calculator. Must have at least 25% chance of prostate cancer development as assessed by the prostate cancer risk calculator.
2. During time of study period, patients must agree not to take any new vitamin supplementation, soy or herbal supplement.
3. Must not be receiving concurrent chemotherapy, radiation or hormonal therapy.
4. No history of prior allergy and intolerability to soy-based products.
5. Must not have been taking any soy supplementation, soy isoflavones or finasteride within 90 days prior to study enrollment.
6. Must be able to safely be on study supplements for period of at least four months.
7. All patients must have been informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
8. All patients must be willing to undergo prestudy and follow-up assessment, including prostate biopsies.

Exclusion Criteria:

1. Patients diagnosed with prostate cancer on initial biopsy
2. Patients with any active malignancy
3. Receiving any concurrent chemotherapy, hormonal therapy or radiation
4. Patient not compliant with treatment for at least 4 months
5. Patients with history of deep vein thrombosis, myocardial infarction, coronary artery disease,and cerebrovascular accident in the last 6 months will also be excluded.
6. Patients on active anticoagulation will be excluded.
7. Patients with liver function tests more than 2 levels of upper limit of normal
8. Patients who develop more than grade 2 toxicity will also be removed from the study

Ages: 55 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Biomarkers will be identified to help predict future prostate cancer risks and patients likely to benefit from preventive strategies | 2 years from completion of enrollment

SECONDARY OUTCOMES:
provide a platform ongoing evaluation of novel preventive agents | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Van Veldhuizen, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Veterans Administration Medical Centenr, Kansas City, Missouri